CLINICAL TRIAL: NCT02854969
Title: Randomized, Cross-over, Open, Unicentric Trial Evaluating Satisfaction With the Use of a Medical Device for the Epinephrine Auto-injector in Patients With Anaphylaxis
Brief Title: Satisfaction of Patient With Anaphylaxis in the Use of a Medical Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adan Medical Innovation, SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AnapphylaxisQoL
Record Dates: First submitted 2016-07-22; First posted 2016-08-04 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2016-08

CONDITIONS: Anaphylaxis
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- epinephrine auto-injector (No Intervention): 3 months using the epinephrine auto-injector alone, and after that 3 more months using the epinephrine auto-injector + medical device
- epinephrine auto-injector + medical device (Experimental): Device: Anapphylaxis is a medical device with a case for an epinephrine autoinjector that connects via Bluetooth to a mobile application
  3 months using the epinephrine auto-injector + medical device , and after that 3 more months using the epinephrine auto-injector alone
  Interventions: Behavioral: Device: Anapphylaxis

INTERVENTIONS:
Behavioral: Device: Anapphylaxis
  Arms: epinephrine auto-injector + medical device

SUMMARY:
Through several questionaries the investigators will measure the satisfaction of patients diagnosed with anaphylaxis in the use of a medical device for the adrenaline autoinjector, a smart case for an epinephrine autoinjector connected via Bluetooth to a mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or above
* Patients diagnosed with Anaphylaxis and an epinephrine auto-injector prescribed
* Patients with a smartphone
* Patients who signed the informed consent

Exclusion Criteria:

* Patients who have not signed the informed consent
* Patients with some limitations for understanding or following correctly the trial procedures
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction through a questionnaire in the use of the medical device | 3 months

SECONDARY OUTCOMES:
Medical device safety | 3 months
  Adverse events related to the medical device
Patient Adherence to the medical device through a questionnaire | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain